CLINICAL TRIAL: NCT06744361
Title: KETamine Sedation As Neuroprotective Agent Following Out-of-hospital Cardiac Arrest (OHCA) - the KETOHCA Trial
Brief Title: Ketamine Sedation As Neuroprotective Agent Following Out-of-hospital Cardiac Arrest
Acronym: KETOHCA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Hassager (Other)
Responsible Party: Sponsor-Investigator, Christian Hassager, Chief Physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-515987-29-00; 2024-515987-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-06; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA)
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-ketamin (Experimental): Intravenous or intraosseous bolus administration at a minimum of 0.5 mg/kg of esketamine
  Interventions: Drug: esketamine hydrochloride
- Propofol (Active Comparator): Prehospital intravenous or intraosseous bolus administration of a minimum dose of 0.25 mg/kg propofol
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: esketamine hydrochloride — Prehospital intravenous or intraosseous bolus administration at a minimum of 0.5 mg/kg of esketamine
  Arms: S-ketamin
Drug: propofol — Prehospital intravenous or intraosseous bolus administration at a minimum dose of 0.25 mg/kg propofol
  Arms: Propofol

SUMMARY:
OHCA is a critical medical emergency with significant mortality and morbidity primarily due to hypoxic-ischemic brain injury (HIBI). Despite advances in resuscitation techniques, the neurological outcomes for survivors remain poor. Current post-resuscitation practices lack specific neuroprotective strategies. Ketamine, an N-Methyl-D-Aspartate (NMDA) receptor antagonist, has shown potential neuroprotective properties in preclinical and clinical studies due to its ability to inhibit excitotoxicity and reduce neuronal apoptosis. This trial hypothesizes that ketamine, when used for sedation in OHCA patients, may offer superior neuroprotective benefits compared to the commonly used sedative propofol. By comparing the effects of ketamine and propofol on neuronal damage markers and long-term neurological outcomes, this study aims to identify a potentially effective intervention to improve the prognosis of OHCA patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years) AND
* resuscitated OHCA of presumed cardiac cause with a shockable first recorded heart rhythm AND
* mean arterial pressure (MAP) >40 mmHg AND
* a decision to perform prehospital intubation.

Exclusion Criteria:

* Advanced life support termination-of-resuscitation (TOR) criteria met
* Systolic blood pressure >190 mmHg
* Known allergy to ketamine or propofol
* Chronic diseases making 180-day survival unlikely
* Body temperature <30° C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Neuron-specific enolase (NSE) measured 48 hours after OHCA | 48 hours after OHCA
  To determine the neuroprotective efficacy of ketamine compared with propofol administered as part of sedation for intubation after initial resuscitation from OHCA

SECONDARY OUTCOMES:
Death from any cause | 180 days after cardiac arrest
  Death from any cause 180 days after cardiac arrest
Neurological outcome: modified Rankin Score (mRS) | At 2 weeks (at discharge)
  Neurological outcome by and modified Rankin Score (mRS). Meassured from 0 to 6, where 0 is no symptoms.
Neurological outcome: Cerebral Performance Categories (CPC) | At 2 weeks (at discharge)
  Neurological outcome by Cerebral Performance Categories (CPC) meassured fra 1-5 (a score of 1 is normal/good cerebral function).
Neurological outcome: modified Rankin Score (mRS) | At 180 days after OHCA.
  Neurological outcome by and modified Rankin Score (mRS). Meassured from 0 to 6, where 0 is no symptoms.
Neurological outcome: modified Rankin Score (mRS) | At 240 days after OHCA.
  Neurological outcome by and modified Rankin Score (mRS). Meassured from 0 to 6, where 0 is no symptoms.
Neurological outcome: Cerebral Performance Categories (CPC) | At 180 days after OHCA.
  Neurological outcome by Cerebral Performance Categories (CPC) meassured fra 1-5 (a score of 1 is normal/good cerebral function).
Neurological outcome: Cerebral Performance Categories (CPC) | At 240 days after OHCA.
  Neurological outcome by Cerebral Performance Categories (CPC) meassured fra 1-5 (a score of 1 is normal/good cerebral function).

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Cardiology, Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense C

IPD SHARING:
Plan to Share IPD: No